CLINICAL TRIAL: NCT06728891
Title: Tumor Deposit at the Fusion Site of the Right Gastric Mesentery and Left Gastric Mesentery in the Patients With Gastric Cancer Who Received Proximal Gastrectomy With D2 Lymphadenectomy Plus Complete Mesogastric Excision for Gastric Cancer: A Prospective Observational Study
Brief Title: Analysis of Tumor Deposit at the Fusion Site of the Right Gastric Mesentery and Left Gastric Mesentery in the Patients With Gastric Cancer Who Received Proximal Gastrectomy
Acronym: zypg001
Status: Recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: 2024-0899-2
Record Dates: First submitted 2024-09-01; First posted 2024-12-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Gastric Carcinoma
Keywords: Gastric cancer; Lymph node dissection; Right gastric mesentery; Tumor deposit
MeSH Terms: conditions — Stomach Neoplasms; Extranodal Extension | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing proximal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision
  Interventions: Other: In addition to routine diagnosis and treatment, no additional intervention measures were taken.

INTERVENTIONS:
Other: In addition to routine diagnosis and treatment, no additional intervention measures were taken. — This study does not impose any intervention on the patients

SUMMARY:
This study aims to evaluate the tumor deposit at the fusion site of the right gastric mesentery and left gastric mesentery in the patients with gastric cancer who received proximal gastrectomy.

DETAILED DESCRIPTION:
In the 6th edition of the Japanese Gastric Cancer Treatment Guidelines; during proximal gastrectomy, D2 lymphadenectomy includes nodes No. 1, No. 2, No. 3a, No. 4sa, No. 4sb, No. 7, No. 8a, No. 9, No. 11p, and No. 11d. When performing D2 surgery for proximal gastric cancer, the dissection typically includes No. 3a (Lymph nodes along the branches of the left gastric artery, including those below the cardia branch) and No. 7 (distributed along the left gastric artery from its root to the bifurcation of the ascending branch), while not including the No. 5 group nodes (located in the upper region of the pylorus between the root of the right gastric artery and the first branch of the gastric wall). In D2 lymphadenectomy plus complete mesogastric excision (CME) for proximal gastric cancer, a complete resection of the left gastric mesentery is performed without removing the right gastric mesentery. However, clinical observations have shown that there may be a fusion between the left and right gastric mesenteries. Merely excising the left gastric mesentery could potentially lead to tumor residue or recurrence in the right mesentery. This study aims to investigate tumor deposit at the fusion site of the right gastric mesentery and left gastric mesentery following D2+CME surgery for proximal gastric cancer, intending to provide evidence-based medical insights for standardizing lymph node clearance in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years
2. Primary gastric adenocarcinoma confirmed by preoperative pathology result
3. cT2-4aN0-3M0 at preoperative evaluation according to the American Joint 8 Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. Patients undergoing proximal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision
5. American Society of Anesthesiologists (ASA) class I, II, or III
6. Written informed consent

Exclusion Criteria:

1. Negative preoperative biopsy
2. Too late tumour stage or metastasis (cT4b/M1)
3. BMI>30 kg/m2
4. previous neoadjuvant chemotherapy or radiotherapy
5. Previous upper abdominal surgery
6. Combined with other malignant diseases
7. Reject operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing proximal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision. At the same time, the patients met the above inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of tumor deposit at the fusion site of the right gastric mesentery and left gastric mesentery; Through postoperative pathological diagnosis | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided